CLINICAL TRIAL: NCT06003010
Title: Efficacy of Perioperative Yoga at Reducing Pain in Surgical AIS Patients
Brief Title: Yoga for Adolescent Idiopathic Scoliosis (AIS) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Pediatric Orthopaedic Society of North America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003670
Record Dates: First submitted 2023-02-16; First posted 2023-08-21 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Adolescent Idiopathic Scoliosis; Spinal Fusion
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (No Intervention): This group will be given standard pre- and post-surgery movement instructions.
- Yoga group (Experimental): This group will be asked to do a 6 week series of yoga videos at home pre- and post-surgery.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — 6 yoga videos to be done 2-3x a week for 6 weeks before and after surgery.
  Arms: Yoga group

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is defined as a three-dimensional lateral deformity of the spine. It is described with a cobb angle of greater than 10 degrees. There is no known etiology of AIS. Once the degrees of curvature become severe (greater than 45 degrees), surgical intervention (posterior spinal fusion - PSF) is often discussed. Most adolescent patients and their families opt for surgical correction to decrease future complications of severe scoliosis, such as decreased vital capacity of the lungs, potential future activity restrictions, cosmetic appearance, and self-esteem. While the patient and family are eager to undergo PSF, they do have concerns. The major concerns are pain control and their ability to return to activities.

In current literature, there are many studies completed regarding pharmacologic pain control management with the use of IV patient-controlled analgesia (PCA) with opioids, narcotics, non-steroidal anti-inflammatories, muscle relaxers, Tylenol, and gabapentin. However, there is not a well-established multimodal pain management plan for postoperative PSF patients. There is also no current literature discussing nonpharmacologic pain management methods, such as stretching, strengthening and yoga, for patients undergoing PSF. There are multiple studies discussing core stabilization used for helping AIS patients non-operatively. There is no literature discussing the use of nonpharmacologic pain management methods for improved pain control (including decreased use of pharmacologic agents) and quicker return to activities.

The aim of this study is to determine if patients with AIS undergoing PSF require fewer pain medications and have an earlier return to activities if completing a yoga program six weeks prior to their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Scoliosis patients
* English speaking patient and parents

Exclusion Criteria:

* Non idiopathic scoliosis diagnosis
* no access to internet or computer
* non-English speaking parents and/or patient

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Morphine Equivalent Units | 7 weeks
  Number of narcotics taken after surgery
Time to first ambulation | 1 week
  How long it takes patient to walk after surgery
Length of hospital stay | 1 week
  How long before the patient was discharged after surgery
Return to school/activities | 7 weeks
  How long before the patient returned to school/activities after surgery
Pain scores | 14 weeks
  Pain scores before and various times after surgery using Faces Pain Scale-Revised. Range is from 0-10. 10 being most severe pain.

SECONDARY OUTCOMES:
Compliance with yoga videos | 14 weeks
  How often patients did yoga videos via patient recorded log and YouTube Analytics

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Children's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All participants will be assigned a study number. Any identifiable information will be stored separately from study data and will only be accessed by authorized team members.